CLINICAL TRIAL: NCT06394115
Title: Assessment of Novel Technology to Facilitate Drainage in Ostomy Pouches: OUTFLOW Study
Acronym: OUTFLOW
Status: Completed | Type: Observational
Sponsor: ConvaTec Inc. (Industry)
Collaborators: Princeton Consumer Research (Other)
Responsible Party: Sponsor
Other Study IDs: OC-21-419
Record Dates: First submitted 2022-07-22; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Colostomy Stoma; Ileostomy - Stoma
Keywords: Ileostomy; Colostomy; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ostomy pouch — Ostomy pouch coated with novel technology

SUMMARY:
The overall aim of this study is to determine the performance and safety of a novel coated material inside Convatec Ostomy Pouches, and to explore the clinical and quality of life benefits that may occur with the use of the test product. A minimum of 30 subjects, and a maximum of 40 subjects will be recruited to obtain 30 complete datasets comprised of a minimum of 15 colostomy and minimum of 10 ileostomies.

ELIGIBILITY:
Inclusion Criteria:

* • Subjects with a colostomy or ileostomy

  * Age 18 years and over
  * Medically stable in the opinion of the investigator
  * Are able and willing to provide informed consent
  * Are able and willing to attend study visits
  * Currently use the same models of pouches as required by the study
  * Have a recent history of frequent pancaking (colostomy patients only)
  * Willing to stop using any lubricants in the pouches whilst participating in the study.
  * Subject has a valid email address for the Investigator to send links to study questionnaires and has access to a web enabled device.

Exclusion Criteria:

* • Subjects with any peristomal skin condition classified as non-intact skin at the time of enrolment

  * Subjects who maybe receiving any concomitant treatment and/or medications which could impact the consistency of effluent during the study period.
  * Allergic to any components of the Novel Lubricant inclusive of Soyabean and/or Vitamin E.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A minimum of 15 colostomy and minimum of 10 ileostomies
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Performance of Convatec ostomy pouches which have the novel coating | 16 days
  To demonstrate the performance of Convatec ostomy pouches which have the novel coating

SECONDARY OUTCOMES:
to investigate the safety of Convatec Ostomy Pouches modified with a novel coating | 16 days
  Evaluation of device related safety events during the treatment period and Evaluation of quality of life and patient perception of product.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Princeton Consumer Research, St. Petersburg, Florida
  - Princeton Consumer Research, Raritan, New Jersey

IPD SHARING:
Plan to Share IPD: No